CLINICAL TRIAL: NCT02165111
Title: A Randomized, Double-Blinded, Placebo-Controlled Clinical Trial Assessing the Therapeutic Efficacy of Botulinum Toxin In Treating Scleroderma-Associated Raynaud's Syndrome
Brief Title: Efficacy of Botulinum Toxin In Scleroderma-Associated Raynaud's Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Scott D. Lifchez, Associate Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA_00087346
Record Dates: First submitted 2014-06-11; First posted 2014-06-17 (Estimated); Results first posted 2016-12-22 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-10

CONDITIONS: Scleroderma; Raynaud's Syndrome
Keywords: Scleroderma, Systemic; Raynaud Disease; Botulinum Toxins, Type A
MeSH Terms: conditions — Scleroderma, Diffuse; Raynaud Disease; Scleroderma, Systemic | interventions — Botulinum Toxins, Type A; Botulinum Toxins; abobotulinumtoxinA; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Onabotulinumtoxin A (Experimental): One hand of each patient will be randomly selected for injection of Botulinum Toxin A (Onabotulinumtoxin A, 20 units/mL).
  Injections are performed using a 30 gauge insulin syringe through the dorsal surface in seven locations: adjacent to the 2nd, 3rd, and 4th common digital arteries through the web spaces (10 units each=0.5mL each), and the radial side of the index finger metacarpal head, the ulnar side of the small finger metacarpal head, and each side of the thumb metacarpal head (5 units each= 0.25mL each). Total treatment dose of Botulinum Toxin A will not exceed 50 units per hand.
  Interventions: Drug: Onabotulinumtoxin A
- Placebo (Placebo Comparator): One hand of each patient will be randomly selected for injection of sterile saline solution (placebo).
  Injections are performed using a 30 gauge insulin syringe through the dorsal surface in seven locations: adjacent to the 2nd, 3rd, and 4th common digital arteries through the web spaces (0.5 mL each), and the radial side of the index finger metacarpal head, the ulnar side of the small finger metacarpal head, and each side of the thumb metacarpal head (0.25 mL each).
  Interventions: Drug: sterile saline solution

INTERVENTIONS:
Drug: Onabotulinumtoxin A
  Other Names: Botox; Botulinum toxin; Dysport
  Arms: Onabotulinumtoxin A
Drug: sterile saline solution
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This is a randomized, double-blinded, clinical trial assessing the therapeutic efficacy of Botulinum toxin A (Onabotulinumtoxin A) in treating scleroderma-associated Raynaud's syndrome. Each patient will undergo injection with a treatment dose of Botulinum toxin A in one randomly-selected hand, and the contralateral hand will be injected with sterile saline (placebo) to serve as a control.

Study participants at the first study visit will complete study questionnaires, their hands will be assessed clinically for digital ulceration, and their hands will undergo non-invasive laser Doppler imaging to assess blood flow. After this initial assessment, the patients will undergo peri-arterial injection of Botulinum toxin A in one hand, and of sterile saline solution (placebo) in the other, in a randomized, blinded manner.

Patient will report the severity of their Raynaud's symptoms weekly over the four month study period. At one month post-injection, the patient will complete study questionnaires, their hands will be assessed clinically for digital ulceration, and their hands will undergo non-invasive laser Doppler imaging. At four months post-injection, the patient will again complete study questionnaires, their hands will be assessed clinically for digital ulceration, and their hands will undergo non-invasive laser Doppler imaging. In addition, patient will be given the option of one week post-injection visit, at which point the same assessment will be performed.

At the conclusion of the study, unblinding will occur.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* Diagnosed with scleroderma.
* Symptoms of Raynaud's syndrome affecting both hands (not necessarily to equal extents)
* Ability to return/be available for follow-up evaluations
* Able and willing to give informed consent
* Able to speak and read in the English language.

Exclusion Criteria:

* A history of Myasthenia gravis.
* Reported allergy or hypersensitivity to any Botulinum toxin preparation.
* Active infection in either hand.
* Patients who have ever received Botulinum toxin vaccine.
* Pregnant or lactating women.
* Females unable or unwilling to maintain abstinence or use contraception for 28 days following the injections.
* Patients who have previously undergone any vascular surgery on the upper extremity, including surgical sympathectomies.
* Current use of any aminoglycoside antibiotic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Lifchez, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Iorio ML, Masden DL, Higgins JP. Botulinum toxin A treatment of Raynaud's phenomenon: a review. Semin Arthritis Rheum. 2012 Feb;41(4):599-603. doi: 10.1016/j.semarthrit.2011.07.006. Epub 2011 Aug 24. PMID 21868066
- [Derived] Bello RJ, Cooney CM, Melamed E, Follmar K, Yenokyan G, Leatherman G, Shah AA, Wigley FM, Hummers LK, Lifchez SD. The Therapeutic Efficacy of Botulinum Toxin in Treating Scleroderma-Associated Raynaud's Phenomenon: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial. Arthritis Rheumatol. 2017 Aug;69(8):1661-1669. doi: 10.1002/art.40123. Epub 2017 Jun 26. PMID 28426903

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Hands
Groups:
- Onabotulinumtoxin A: One hand of each patient was randomly selected for injection of Botulinum Toxin A (Onabotulinumtoxin A, 20 units/mL).
  Injections were performed using a 30 gauge insulin syringe through the dorsal surface in seven locations: adjacent to the 2nd, 3rd, and 4th common digital arteries through the web spaces (10 units each=0.5mL each), and the radial side of the index finger metacarpal head, the ulnar side of the small finger metacarpal head, and each side of the thumb metacarpal head (5 units each= 0.25mL each). Total treatment dose of Botulinum Toxin A will not exceed 50 units per hand.
- Placebo: One hand of each patient was randomly selected for injection of sterile saline solution (placebo).
  Injections were performed using a 30 gauge insulin syringe through the dorsal surface in seven locations: adjacent to the 2nd, 3rd, and 4th common digital arteries through the web spaces (0.5 mL each), and the radial side of the index finger metacarpal head, the ulnar side of the small finger metacarpal head, and each side of the thumb metacarpal head (0.25 mL each).
Period: Overall Study
Arm/Group | Onabotulinumtoxin A | Placebo
Started | 40; 40 Hands | 40; 40 Hands
Completed | 40; 40 Hands | 40; 40 Hands
Not Completed | 0; 0 Hands | 0; 0 Hands

BASELINE CHARACTERISTICS:
Population: This trial was designed as a within-participant study where one of the 40 participants' hands was randomized to receive Onabotulinumtoxin A and the other to receive placebo. Each participant thus contributed two hands to the total number of units analyzed.
Units Other Than Participants: Hands
Groups:
- Onabotulinumtoxin A: One hand of each patient was be randomly selected for injection of Botulinum Toxin A (Onabotulinumtoxin A, 20 units/mL).
  Injections were performed using a 30 gauge insulin syringe through the dorsal surface in seven locations: adjacent to the 2nd, 3rd, and 4th common digital arteries through the web spaces (10 units each=0.5mL each), and the radial side of the index finger metacarpal head, the ulnar side of the small finger metacarpal head, and each side of the thumb metacarpal head (5 units each= 0.25mL each). Total treatment dose of Botulinum Toxin A will not exceed 50 units per hand.
  Onabotulinumtoxin A
- Placebo: One hand of each patient was randomly selected for injection of sterile saline solution (placebo).
  Injections were performed using a 30 gauge insulin syringe through the dorsal surface in seven locations: adjacent to the 2nd, 3rd, and 4th common digital arteries through the web spaces (0.5 mL each), and the radial side of the index finger metacarpal head, the ulnar side of the small finger metacarpal head, and each side of the thumb metacarpal head (0.25 mL each).
  sterile saline solution
- Total: Total of all reporting groups
Arm/Group | Onabotulinumtoxin A | Placebo | Total
Number analyzed (Participants) | 40 | 40 | 40
Number analyzed (Hands) | 40 | 40 | 80
Age, Categorical [Count of Units; unit: Hands]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 35 | 70
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (12.33) | 51.9 (12.33) | 51.9 (12.33)
Gender [Count of Units; unit: Hands]
  Female | 9 | 9 | 18
  Male | 31 | 31 | 62
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 40
Laser Doppler Imaging Blood Flow [Mean (Standard Deviation); unit: LDI flux units] — Laser Doppler Imaging measures blood flow using a low-energy laser beam that quantifies the Doppler effect between red blood cells and a scanner to determine blood flow speed, allowing non-invasive, objective measurement of superficial cutaneous blood flow.
  LDI flux units | 398.24 (190.27) | 395.65 (189.17) | 396.94 (188.52)

OUTCOME MEASURES:

1. Primary Outcome: Change in Digital Blood Flow From Pre- to Post-injection.
Description: The primary outcome measure is change in blood flow to the fingers, from a pre-injection baseline to post-injection follow-up visit as measured by non-invasive laser Doppler imaging.
Time Frame: Measured pre-injection and at one month post-injection.
Measure: Mean (95% Confidence Interval); unit: Blood flow, measured in LDI flux units,
Groups:
- Onabotulinumtoxin A: One hand of each patient was randomly selected for injection of Botulinum Toxin A (Onabotulinumtoxin A, 20 units/mL).
  Injections were performed using a 30 gauge insulin syringe through the dorsal surface in seven locations: adjacent to the 2nd, 3rd, and 4th common digital arteries through the web spaces (10 units each=0.5mL each), and the radial side of the index finger metacarpal head, the ulnar side of the small finger metacarpal head, and each side of the thumb metacarpal head (5 units each= 0.25mL each). Total treatment dose of Botulinum Toxin A will not exceed 50 units per hand.
  Onabotulinumtoxin A
Arm/Group | Onabotulinumtoxin A | Placebo
Number analyzed (Participants) | 40 | 40
Blood flow, measured in LDI flux units, | -36.19 [-78.49 to 6.12] | -6.10 [-46.28 to 34.07]

2. Secondary Outcome: Rate of Change in Raynaud's Phenomenon Symptoms Measured With the Raynaud's Condition Score.
Description: Raynaud's Condition Score is a patient-reported, validated outcomes scale that measures the severity of Raynaud's phenomenon on a scale of 0 ("No difficulty") to 10 ("Extreme difficulty"), where higher values represent a worse outcome.
  Data from each weekly report were combined using a statistical model (generalized linear population-average model) to calculate a weekly rate of change for each participant's hand, where a negative value represents a improvement over time and a positive value represents worsening over time.
Time Frame: Weekly rate of change over the four-month study period.
Measure: Mean (95% Confidence Interval); unit: change in RCS/week
Groups:
- Onabotulinumtoxin A: One hand of each patient were randomly selected for injection of Botulinum Toxin A (Onabotulinumtoxin A, 20 units/mL).
  Injections were performed using a 30 gauge insulin syringe through the dorsal surface in seven locations: adjacent to the 2nd, 3rd, and 4th common digital arteries through the web spaces (10 units each=0.5mL each), and the radial side of the index finger metacarpal head, the ulnar side of the small finger metacarpal head, and each side of the thumb metacarpal head (5 units each= 0.25mL each). Total treatment dose of Botulinum Toxin A will not exceed 50 units per hand.
  Onabotulinumtoxin A
- Placebo: One hand of each patient were randomly selected for injection of sterile saline solution (placebo).
  Injections were performed using a 30 gauge insulin syringe through the dorsal surface in seven locations: adjacent to the 2nd, 3rd, and 4th common digital arteries through the web spaces (0.5 mL each), and the radial side of the index finger metacarpal head, the ulnar side of the small finger metacarpal head, and each side of the thumb metacarpal head (0.25 mL each).
  sterile saline solution
Arm/Group | Onabotulinumtoxin A | Placebo
Number analyzed (Participants) | 40 | 40
change in RCS/week | -0.18 [-0.22 to -0.13] | -0.14 [-0.18 to -0.11]

3. Secondary Outcome: Number of Ulcers as Measure of Digital Ulcer Healing
Description: A secondary outcome of this study is the number of digital ulcers as determined by clinical examination. Mean number of ulcers was calculated as total number of ulcers / total number of hands in each group.
Time Frame: Measured at one month post-injection.
Measure: Mean (Standard Deviation); unit: Number of ulcers
Arm/Group | Onabotulinumtoxin A | Placebo
Number analyzed (Participants) | 40 | 40
Number of ulcers | 0.45 (0.90) | 0.53 (0.93)

4. Secondary Outcome: Assessment of Raynaud's Symptoms Severity Using the Quick-DASH Score.
Description: A secondary outcome of this study is severity of Raynaud's symptoms as measured by the self-reported Quick-DASH score. The Quick-DASH scores measures the degree of hand and upper extremity function on a scale of 0 (not limited) to 100 (severely limited) where a higher value represents a worse outcome.
Time Frame: Measured at one month post-injection.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Onabotulinumtoxin A | Placebo
Number analyzed (Participants) | 40 | 40
Units on a scale | 26.96 (20.68) | 29.11 (23.80)

5. Secondary Outcome: Assessment of Raynaud's Symptom Severity Using the McCabe Cold Sensitivity Score.
Description: A secondary outcome of this study is the patient-reported sensitivity to coldness as measured by the McCabe Cold Sensitivity score. Patients' answers on this validated instrument are scored on a scale from 0 (no sensitivity) to 400 (extreme sensitivity), where a higher number represents a worse outcome.
Time Frame: Measured at one month post-injection.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Onabotulinumtoxin A | Placebo
Number analyzed (Participants) | 40 | 40
Units on a scale | 185.31 (74.19) | 187.19 (86.76)

6. Secondary Outcome: Assessment of Raynaud's Symptom Severity Using the VAS for Pain.
Description: A secondary outcome of this study is pain as measured by the validated visual-analog scale (VAS) for pain. The VAS pain instrument measures pain on a scale from 0 cm (no pain) to 10 cm (extreme pain)
Time Frame: Measured at one month post-injection.
Measure: Mean (Standard Deviation); unit: centimeters measured on a visual scale
Arm/Group | Onabotulinumtoxin A | Placebo
Number analyzed (Participants) | 40 | 40
centimeters measured on a visual scale | 2.68 (2.57) | 3.05 (2.77)

ADVERSE EVENTS:
Time Frame: 4 months
Description: Participants were asked about adverse events during a safety call at 1 week post-injection and in-person visits at 1-month and 4-months post-injection visits.
Arm/Group | Onabotulinumtoxin A | Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 2/40 | 0/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Onabotulinumtoxin A (N=40) | Placebo (N=40)
Intrinsic muscle weakness (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Multi-level data prevents conclusions from being drawn from aggregate data alone. High degree of variability of the results suggests a heterogeneous group of scleroderma patients. Screening methods and no dose escalation may explain negative findings

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No